CLINICAL TRIAL: NCT02944981
Title: Gabapentin Premedication to Reduce Postoperative Nausea and Vomiting in Surgical Patient Receiving Spinal Morphine
Brief Title: Gabapentin to Reduce Postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HE571129
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Gabapentin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental): Patient receiving oral gabapentin 600 mg preoperatively
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Patient receiving oral placebo tablet preoperatively
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Single oral dose
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo — Single oral dose
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The intrathecal administration of morphine is gaining popularity. It is easy to do and can reduce the pain after surgery up to 24 hours. However, it causes postoperative nausea and vomiting more than other methods providing postoperative analgesia. Patients suffering from these side effects have to spend a longer period of time recovering in the hospital with high cost of medical treatment.

DETAILED DESCRIPTION:
Objective: to study the efficacy of oral administrating of gabapentin 600 mg before surgery to reduce the postoperative nausea and vomiting in patients receiving intrathecal morphine.

Methods: Eighty patients undergoing orthopedic surgery and receiving intrathecal morphine will be randomized into 2 groups. The first group will receive oral gabapentin 600 mg and the second group will receive a placebo tablet. Both groups will receive a standard prophylactic medication for postoperative nausea and vomiting. The degrees of nausea and vomiting in both groups will be assessed over 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general or regional anesthesia receiving spinal morphine
* ASA physical status I-III

Exclusion Criteria:

* Patients with allergy to morphine or gabapentin
* Chronic use of narcotics
* Psychotic
* Bleeding disorder
* Cardiovascular disorder
* Liver or renal failure
* Pregnancy or breast feeding
* Neurologic disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting (grade 1-3) | through study completion, an average of 24 hours
  PONV grading: 0 = none; 1 = mild; 2 = moderate; 3 = severe

CONTACTS AND LOCATIONS:
Overall Officials: Sirirat Tribuddharat, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand
Locations (1):
- Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dahl JB, Jeppesen IS, Jorgensen H, Wetterslev J, Moiniche S. Intraoperative and postoperative analgesic efficacy and adverse effects of intrathecal opioids in patients undergoing cesarean section with spinal anesthesia: a qualitative and quantitative systematic review of randomized controlled trials. Anesthesiology. 1999 Dec;91(6):1919-27. doi: 10.1097/00000542-199912000-00045. No abstract available. PMID 10598635
- [Result] Devys JM, Mora A, Plaud B, Jayr C, Laplanche A, Raynard B, Lasser P, Debaene B. Intrathecal + PCA morphine improves analgesia during the first 24 hr after major abdominal surgery compared to PCA alone. Can J Anaesth. 2003 Apr;50(4):355-61. doi: 10.1007/BF03021032. English, French. PMID 12670812
- [Result] Pandey CK, Priye S, Ambesh SP, Singh S, Singh U, Singh PK. Prophylactic gabapentin for prevention of postoperative nausea and vomiting in patients undergoing laparoscopic cholecystectomy: a randomized, double-blind, placebo-controlled study. J Postgrad Med. 2006 Apr-Jun;52(2):97-100. PMID 16679671
- [Result] Rorarius MG, Mennander S, Suominen P, Rintala S, Puura A, Pirhonen R, Salmelin R, Haanpaa M, Kujansuu E, Yli-Hankala A. Gabapentin for the prevention of postoperative pain after vaginal hysterectomy. Pain. 2004 Jul;110(1-2):175-81. doi: 10.1016/j.pain.2004.03.023. PMID 15275765